CLINICAL TRIAL: NCT05766969
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Using Cannabidiol and Palmitoylethanolamide for the Treatment of Painful Diabetic Peripheral Neuropathy of the Feet
Brief Title: Diabetic Neuropathic Pain Relief, 6 Weeks Dosage Sublingual Water-soluble CBD/PEA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pure Green Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The DIA/NPR-6 Study
Record Dates: First submitted 2023-03-02; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Intervention Model Description: There are 2 groups in this trial: interventional group (active drug) and control group (placebo).
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized at a 2:1 ratio.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD/PEA (Experimental): Subject will receive a 42-day supply of 10/50 mg CBD/PEA sublingual tablets to be taken 3 times a day for 42 days.
  Interventions: Drug: CBD/PEA
- Placebo Control (Placebo Comparator): A placebo sublingual tablet to be taken three times a day for 42 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD/PEA — A water-soluble sublingual tablet containing 10/50 mg of CBD/PEA.
  Other Names: PGP-DPN-10/50
  Arms: CBD/PEA
Drug: Placebo — An inactive compound.
  Arms: Placebo Control

SUMMARY:
The purpose of the study is to evaluate whether the DIA/NPR-6 is a better pain reliever in patients with diabetic neuropathic pain of the feet compared to placebo.

DETAILED DESCRIPTION:
Subjects will be enrolled in the study for a maximum of 63 days, including an optional 14-day screening period, 42 days of active product administration, and followed by post-treatment blood work, EKG, and questionnaires within 24-hours following study treatment completion and a psychiatric and primary health care provider evaluation within 1 week of trial completion.

The primary objective of this study is:

* To evaluate the impact of PGP-010-50-1 on subject's painful diabetic neuropathic pain (pDNP), anxiety, and sleep quality compared to a placebo control.
* To evaluate the impact of PGP-010-50-1 on the subject's impression of their response to the treatment compared to a placebo control.

The secondary objectives of this study are:

* To evaluate the safety of PGP-010-50-1 for the treatment of painful diabetic peripheral neuropathy (DPN) of the feet compared to a placebo control
* To evaluate PGP-010-50-1 on liver function.
* To evaluate PGP-010-50-1 on Hbg A1C

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 21 years of age.
2. Subject is or under the age of 65 years of age.
3. Subject has a primary health care provider and gives permission for PG Pharma to contact the primary health care provider.
4. Subject has a diagnosis of diabetic neuropathic pain of the feet .
5. Subject has a mean pain scale score of ≥ 4 and ≤ 8 recorded localized to the foot in the 7 days prior to randomization.
6. If female, the subject is postmenopausal (> 1 year), surgically sterile (> 3 months), had a hysterectomy, or is currently using 2 effective forms of birth control.
7. Subject has not taken marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 14 days prior to this study, and agrees to not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study.
8. Subject is willing to provide his/her written informed consent to participate in the study as stated in the informed consent document.
9. Subject has a smart phone, knows how to use it, and is willing to use it for accessing and interacting with an electronic diary to enter trial information for the duration of the study - 57 days. (up to 14-day screening period and 42 days active dosing and 1 day post dosing.

Exclusion Criteria:

1. Subject is pregnant or lactating.
2. Subject is unwilling to utilize two forms of birth control with partner.
3. Male subject is unwilling to agree to not donate sperm from the time of dosing until 90 days after dosing of study drug.
4. Subject has an allergy to cannabis, the Cannabaceae plant family (e.g., hemp, hops), palmitoylethanolamide, or terpenes.
5. Subject has a known allergy to active or inert ingredients of the investigational product.
6. Subject is taking a concomitant medication or treatment that would complicate use or interpretation of the study drug's effects (examples include: Cannabis or any cannabinoid products; Any drug or herbal product that influences the endocannabinoid system (ECS)). However, subjects are allowed to continue gabapentin and pregabalin medications, if the subject still meets the pain scale inclusion criteria, evidencing lack of effectiveness of their concomitant pain medication.
7. Subjects on SNRIs or SSRIs.
8. Subject is taking marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 14 days prior to this study, and does not promise that they will not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study;
9. Subject has shortness of breath.
10. Subject has uncontrolled asthma.
11. Subject has a fever and/or productive cough.
12. Subject has unstable angina, uncontrolled hypertension.
13. Subject currently or has a history of congestive heart failure.
14. Subject meets any DSM-V criteria for current, major psychiatric illness, including but not limited to: bipolar disorder, major depressive disorder, psychosis, or substance abuse disorder.
15. Subject has a personal or family history of schizophrenia.
16. Subject has a personal history or currently has suicidal ideation or attempted suicide.
17. Subject has a major neurological disorder, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, history of traumatic brain injury/head injury, and seizures.
18. Subject has a history of multiple sclerosis.
19. Subject is currently taking any form of opioids.
20. Subject has a history of substance or alcohol abuse.
21. Subject has clinically significant illness, including cardiovascular disorders.
22. Subject has any condition in which the investigator believes will confound the data of the study or could put the subject at risk of harm.
23. Subject does not have access to a smart phone or does not know how to use a smart phone application.
24. Subject is not within 30 miles of a Quest Diagnostics laboratory.
25. The skin under the tongue or anywhere in the oral cavity is not intact.
26. Subject has abnormal liver function test results.
27. Subject has a history of abnormal liver dysfunction or liver pathology.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2023-12-05 (Estimated); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
Pain as assessed by Numerical Pain Rating Scale (NPRS) | Six Weeks
  To evaluate the impact of DIA/NPR-6 on the subject's neuropathic pain as assessed by utilizing a Numeric Pain Rating Scale (NPRS). NPRS is from 0-10, where higher scores indicate worse pain, and lower scores indicate less pain reported by the subject.
Pain as measured by the Brief Pain Inventory (BPI) | Six Weeks
  To evaluate the impact of DIA/NPR-6 on the subject's neuropathic pain as assessed by utilizing a Brief Pain Inventory (BPI) where patients will answer 15 questions regarding their pain.
Anxiety as measured by the Self-Rating Anxiety Scale (SAS) | Six Weeks
  To evaluate the impact of DIA/NPR-6 on the subject's anxiety as assessed by the Self-Rating Anxiety Scale (SAS). Subjects will complete SAS prior to first dose and during post-treatment.
Sleep as measured by the Pittsburg Sleep Quality Index (PSQI) | Six Weeks
  To evaluate the impact of DIA/NPR-6 on the subject's sleep as assessed by the Pittsburgh Sleep Quality Index (PSQI). Subjects will be evaluated pre- and post-treatment. The PSQI produces a global score and 6 subscales, Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbances, Use of Sleeping Medications, and Daytime Dysfunction.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events as assessed by CTCAE v4.0 | Six Weeks
  To evaluate the safety of DIA/NPR-6 for the treatment of painful DPN of the feet compared to a placebo control assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Subject's Response to Treatment as assessed by Patient's Global Impression of Change (PGIC) | Six Weeks
  To evaluate the impact of DIA/NPR-6 on the subject's impression of their response to the treatment compared to a placebo control as assessed by Patient's Global Impression of Change (PGIC). Subjects indicate their overall impression of their response to treatment on 0-10 scale, where a higher number represents the subject feeling worse than before the intervention, and a lower number represents the subject feeling better than before the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kimless, MD, Principal Investigator — Pure Green Pharmaceuticals Inc.
Locations (1):
- Pure Green Pharmaceuticals Inc., Southfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quattrini C, Tesfaye S. Understanding the impact of painful diabetic neuropathy. Diabetes Metab Res Rev. 2003 Jan-Feb;19 Suppl 1:S2-8. doi: 10.1002/dmrr.360. PMID 12577252
- [Background] Callaghan BC, Cheng HT, Stables CL, Smith AL, Feldman EL. Diabetic neuropathy: clinical manifestations and current treatments. Lancet Neurol. 2012 Jun;11(6):521-34. doi: 10.1016/S1474-4422(12)70065-0. Epub 2012 May 16. PMID 22608666
- [Background] Argoff CE, Cole BE, Fishbain DA, Irving GA. Diabetic peripheral neuropathic pain: clinical and quality-of-life issues. Mayo Clin Proc. 2006 Apr;81(4 Suppl):S3-11. doi: 10.1016/s0025-6196(11)61474-2. PMID 16608048
- [Background] Sadosky A, Mardekian J, Parsons B, Hopps M, Bienen EJ, Markman J. Healthcare utilization and costs in diabetes relative to the clinical spectrum of painful diabetic peripheral neuropathy. J Diabetes Complications. 2015 Mar;29(2):212-7. doi: 10.1016/j.jdiacomp.2014.10.013. Epub 2014 Nov 8. PMID 25498300
- [Background] Gordois A, Scuffham P, Shearer A, Oglesby A, Tobian JA. The health care costs of diabetic peripheral neuropathy in the US. Diabetes Care. 2003 Jun;26(6):1790-5. doi: 10.2337/diacare.26.6.1790. PMID 12766111
- [Background] Singh R, Kishore L, Kaur N. Diabetic peripheral neuropathy: current perspective and future directions. Pharmacol Res. 2014 Feb;80:21-35. doi: 10.1016/j.phrs.2013.12.005. Epub 2013 Dec 25. PMID 24373831
- [Background] Wallace MS, Marcotte TD, Umlauf A, Gouaux B, Atkinson JH. Efficacy of Inhaled Cannabis on Painful Diabetic Neuropathy. J Pain. 2015 Jul;16(7):616-27. doi: 10.1016/j.jpain.2015.03.008. Epub 2015 Apr 3. PMID 25843054
- [Background] Bridges D, Ahmad K, Rice AS. The synthetic cannabinoid WIN55,212-2 attenuates hyperalgesia and allodynia in a rat model of neuropathic pain. Br J Pharmacol. 2001 Jun;133(4):586-94. doi: 10.1038/sj.bjp.0704110. PMID 11399676
- [Background] De Vry J, Denzer D, Reissmueller E, Eijckenboom M, Heil M, Meier H, Mauler F. 3-[2-cyano-3-(trifluoromethyl)phenoxy]phenyl-4,4,4-trifluoro-1-butanesulfonate (BAY 59-3074): a novel cannabinoid Cb1/Cb2 receptor partial agonist with antihyperalgesic and antiallodynic effects. J Pharmacol Exp Ther. 2004 Aug;310(2):620-32. doi: 10.1124/jpet.103.062836. Epub 2004 May 12. PMID 15140913
- [Background] Abrams DI, Jay CA, Shade SB, Vizoso H, Reda H, Press S, Kelly ME, Rowbotham MC, Petersen KL. Cannabis in painful HIV-associated sensory neuropathy: a randomized placebo-controlled trial. Neurology. 2007 Feb 13;68(7):515-21. doi: 10.1212/01.wnl.0000253187.66183.9c. PMID 17296917
- [Background] Ware MA, Wang T, Shapiro S, Robinson A, Ducruet T, Huynh T, Gamsa A, Bennett GJ, Collet JP. Smoked cannabis for chronic neuropathic pain: a randomized controlled trial. CMAJ. 2010 Oct 5;182(14):E694-701. doi: 10.1503/cmaj.091414. Epub 2010 Aug 30. PMID 20805210
- [Background] Wilsey B, Marcotte T, Deutsch R, Gouaux B, Sakai S, Donaghe H. Low-dose vaporized cannabis significantly improves neuropathic pain. J Pain. 2013 Feb;14(2):136-48. doi: 10.1016/j.jpain.2012.10.009. Epub 2012 Dec 11. PMID 23237736
- [Background] Wilsey B, Marcotte T, Tsodikov A, Millman J, Bentley H, Gouaux B, Fishman S. A randomized, placebo-controlled, crossover trial of cannabis cigarettes in neuropathic pain. J Pain. 2008 Jun;9(6):506-21. doi: 10.1016/j.jpain.2007.12.010. Epub 2008 Apr 10. PMID 18403272
- [Background] Johnson JR, Burnell-Nugent M, Lossignol D, Ganae-Motan ED, Potts R, Fallon MT. Multicenter, double-blind, randomized, placebo-controlled, parallel-group study of the efficacy, safety, and tolerability of THC:CBD extract and THC extract in patients with intractable cancer-related pain. J Pain Symptom Manage. 2010 Feb;39(2):167-79. doi: 10.1016/j.jpainsymman.2009.06.008. Epub 2009 Nov 5. PMID 19896326
- [Background] De Gregorio D, McLaughlin RJ, Posa L, Ochoa-Sanchez R, Enns J, Lopez-Canul M, Aboud M, Maione S, Comai S, Gobbi G. Cannabidiol modulates serotonergic transmission and reverses both allodynia and anxiety-like behavior in a model of neuropathic pain. Pain. 2019 Jan;160(1):136-150. doi: 10.1097/j.pain.0000000000001386. PMID 30157131